CLINICAL TRIAL: NCT01380379
Title: A Pilot Study of Self-Defense Training in Women With Trauma
Brief Title: Self-Defense Training in Women With Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Senior Research Scholar, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04152011-7701; 20776
Record Dates: First submitted 2011-05-18; First posted 2011-06-27 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Depression; Anxiety; Stress Disorders, Post-Traumatic
Keywords: physical violence; sexual violence
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Life skills and self-defense training (Experimental): Women will participate in a therapeutic group which covers education, skills, and empowerment activities.
  Interventions: Behavioral: Life skills and self-defense training

INTERVENTIONS:
Behavioral: Life skills and self-defense training — 8 week class which meets once per week for 2.5 hours. Each class contains the following components: 1) life skills/education training. This includes basic education about physical and sexual assaults, assault risks, dating and communication, assertiveness training and boundary setting, 2) physical self-defense training, 3) supportive therapy/debriefing.

SUMMARY:
Previous research has shown that self-defense training can lead to gains in women's assertiveness, self-esteem, self-efficacy, and physical competence, and decreases in anxiety, helplessness, fear, and avoidant behaviors. However, most of this research has been conducted with healthy women who had not previously experienced physical or sexual violence. The investigators believe that women with such trauma histories require additional care because of potential triggering symptoms. As such, the investigators are mindful of the potential for triggering trauma symptoms and will work with the women so that they feel safe and comfortable in their participation. This pilot study aims to examine whether similar psychological gains from self-defense training are made in women who have previous experiences of physical and/or sexual violence.

DETAILED DESCRIPTION:
There is a high rate of violence against women in the United States. For example, at least 1 in 6 women will experience an attempted or completed rape in their lifetime (Tjaden & Thoenees, 2000). The high physical, emotional, economic and social costs of such violence are staggering. In particular, there can be a serious impact on mental health, with both immediate and long-term consequences (e.g., Coker et al., 2000). The aim of this project is to examine the psychological benefits of a class, which incorporates psychological and physical self-defense skills, for women who have been the victim of sexual or physical violence.

A small literature suggests that women who take self-defense classes have increases in general self-efficacy and self-esteem (e.g.,Ozer and Bandura, 1990). This project is focusing on women who already have a history of physical or sexual violence. The investigators hypothesize that women who already have such a history of violence will benefit from a self-defense class that incorporates psychoeducation and brief psychology treatments in order to successfully participate in such a class and that ultimately it will improve their psychological well-being.

Potential participants will first do a short phone screening to see whether they may be eligible for the study. If so, they will be brought into the clinic for a full eligibility assessment.

Eligibility Procedures: Before entering the study, participants will participate in an eligibility interview. This will consist of a psychiatric interview (e.g., portions of the SCID and psychiatric rating scales), trauma history (e.g. CAPS), and physical health assessment. Participants will either need approval from their primary care physician to participate in the physical self-defense portion of the study or have a brief physical exam will a physician on the research team.

If the participant is eligible for the study, they will be added to the list of participants. Once an adequate number of participants have been screened and determine eligible for the study, they will participate in the group for 8 weeks.

Participants will fill out a series of questionnaires pre- and post- the course. Each set of questionnaires should take less than 1 hour to complete. In addition, the investigators conducted a 6-month post-class, follow up assessment.

Self-defense class: The self-defense program is an eight week curriculum that meets once per week for 2.5 hours per session. The course which involves three components. The first component is a psycho-educational component which provides current basic information about physical and sexual assaults and also skill building, such as assertiveness, communication skills, and boundary setting. The second component of each class is physical resistance techniques which offers ample training. This includes information about basic targets, punches, and kicks, as well as breaking out of holds and other resistance skills. The third component of each class includes a supportive psychotherapy debriefing session. Following participation in the self-defense class all participants will be required to come for an in-person, debriefing interview.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 21-65 years
2. History of physical and/or sexual violence, with subsequent interpersonal or psychological distress (e.g., depression or anxiety) related to this history.

Exclusion Criteria:

1. Substance abuse in the past 6 months
2. Significant medical conditions that would preclude safe participation in the study
3. High levels of depression with significant suicide risk
4. Pregnant women
5. Active symptoms of psychosis or psychiatric instability
6. History of assaultive behavior or is judged to be at potential risk to assault others.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Life Skills and Self-defense Training
Started | 9
Completed | 8
Not Completed | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Life Skills and Self-defense Training
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.38 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-efficacy From Baseline to Post-treatment
Description: General self-efficacy (Schwartz and Jerusalem, 1993) is a measure of one's perceived self-competence. Scores are summed across 10 items, and range between 10-40, where higher scores reflect a stronger sense of personal competence.
Time Frame: Change in GSE from baseline to 8 weeks
Population: The data is the change in general self efficacy from baseline to post-class, with higher scores indicating a greater increase in self-efficacy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Life Skills and Self-defense Training
Number analyzed (Participants) | 8
units on a scale
  Baseline General Self efficacy | 23.38 (5.8)
  Week 8 (post-class) GSE | 29.63 (3.0)
Statistical Analysis 1: Comparison: Life Skills and Self-defense Training; Test type: Superiority or Other; p < .01, t-test, 2 sided; Single group comparison pre-post change score, compared to a value of 0 (no change)

2. Secondary Outcome: Change in Assertiveness Between Baseline and Post-intervention
Description: Measured by the Rathus Assertiveness Schedule (Rathus, 1973). Rathus Assertiveness Scale is a 30-item scale assessing assertive behavior in a variety of situations. Each item is rated on a 6-point Likert scale from +3 (very characteristic of me) to -3 (very uncharacteristic of me). Total scores range from +90, which is equivalent of very assertive behavior to -90, which is equivalent to very unassertive behavior.
  The positive change indicates an increase in assertive behavior.
Time Frame: Change in assertiveness from baseline to post-class (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Life Skills and Self-defense Training
Number analyzed (Participants) | 8
units on a scale
  Baseline Assertiveness Total | -24.88 (34.6)
  Week 8 (post-class) Assertiveness Total | -15.88 (33.85)
Statistical Analysis 1: Comparison: Life Skills and Self-defense Training; Test type: Superiority or Other; p < .04, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Life Skills and Self-defense Training
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Life Skills and Self-defense Training (N=8)
Dissociation during class (Psychiatric disorders) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No